CLINICAL TRIAL: NCT06502743
Title: Phase 2 Study of First-line Carboplatin and Paclitaxel in Combination With Pembrolizumab, Followed by Maintenance Pembrolizumab With or Without Nesuparib, in Patients With Newly Diagnosed Advanced or Recurrent MMR-proficient (pMMR) Endometrial Cancer
Brief Title: First-line Carboplatin and Paclitaxel in Combination With Pembrolizumab, Followed by Maintenance Pembrolizumab With or Without Nesuparib, in Patients With Newly Diagnosed Advanced or Recurrent MMR-proficient (pMMR) Endometrial Cancer
Acronym: PENELOPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Onconic Therapeutics Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, JUNGYUN LEE, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2024-0577
Record Dates: First submitted 2024-06-23; First posted 2024-07-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer; Recurrent Endometrial Carcinoma; Endometrial Carcinoma; Gynecologycal Cancer; Endometrial Neoplasms
Keywords: Nesuparib; pMMR; MMR-proficient
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part B - Pembrolizumab monotherapy (Experimental): Chemotherapy Treatment Pembrolizumab 200 mg IV Day 1 + Paclitaxel 175mg/m2 IV over 3 hours Day 1 + Carboplatin AUC 5 IV Day 1 x 6 cycles (one cycle = 3 weeks
  Maintenance Treatment Pembrolizumab 400 mg IV Day 1 x up to 14 cycles (o ne cycle = 6 weeks )
  Maximum number of Pembrolizumab cycles (Chemotherapy Treatment + maintenance Treatment ) = 20
  Interventions: Drug: Pembrolizumab
- Part B - Pembrolizumab and nesuparib combination therapy (Experimental): Combination therapy Chemotherapy Treatment Pembrolizumab 200 mg IV Day 1 + Paclitaxel 175mg/m2 IV over 3 hours Day + Carboplatin AUC 5 IV Day 1 x 6 cycles (one cycle = 3 weeks)
  Maintenance Treatment Pembrolizumab 400 mg IV Day 1 + Nesuparib 150mg or 100mg QD PO x up to 14 cycles (o ne cycle = 6 weeks )
  Maximum number of Pembrolizumab cycles (Chemotherapy Treatment + maintenance Treatment ) = 20
  Interventions: Drug: Nesuparib; Drug: Pembrolizumab
- Part A - Safety Run-in Phase (Experimental): Chemotherapy Treatment:
  Pembrolizumab 200 mg IV Day 1 + Paclitaxel 175mg/m2 IV over 3 hours Day 1 + Carboplatin AUC 5 IV Day 1 x 6 cycles (one cycle = 3 weeks)
  Maintenance Treatment:
  Pembrolizumab 400 mg IV Day 1 + Nesuparib 150mg or 100mg QD PO x up to 14 cycles (one cycle = 6 weeks)
  Maximum number of Pembrolizumab cycles (Chemotherapy Treatment + Maintenance Treatment) = 20
  Interventions: Drug: Nesuparib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nesuparib — Nesuparib 150mg or 100mg, QD, PO
  Arms: Part A - Safety Run-in Phase; Part B - Pembrolizumab and nesuparib combination therapy
Drug: Pembrolizumab — Pembrolizumab 400mg, IV, Q6W

SUMMARY:
The goal of this study is listed below.

Part A (Safety Run-in Phase) : To determine feasibility of pembrolizumab and nesuparib combination as maintenance therapy in patients with MMR-proficient advanced and recurrent endometrial cancer. Feasibility is defined as a dose-limiting toxicity (DLT) rate less than or equal to 33%.

Part B (Randomization Phase)

: To evaluate the efficacy of pembrolizumab and nesuparib combination/ pembrolizumab monotherapy as maintenance therapy in patients with MMR-proficient advanced stage and recurrent endometrial cancer. Efficacy will be assessed by investigator assessed progression free survival (PFS) as assessed by RECIST 1.1.

DETAILED DESCRIPTION:
Part A(Safety Run-in Phase) - Pembrolizumab+ paclitaxel+ carboplatin followed by pembrolizumab combination with nesuparib

Part B(Randomization Phase)

- Pembrolizumab+ p aclitaxel+ Carboplatin followed by Pembrolizumab combination with Nesuparib vs Pembrolizumab+ Paclitaxel+ Carboplatin followed by Pembrolizumab monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be female ≥ 19 years of age
2. Histologic confirmation of the original primary tumor is required. Patients with the following histologic types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, carcinosarcoma, adenocarcinoma not otherwise specified (N.O.S.).
3. Measurable stage III, measurable stage IVA, stage IVB (with or without measurable disease) or recurrent (with or without measurable disease) endometrial cancer.
4. MMR proficient confirmed by institutional (local) MMR IHC testing.
5. Patient must provide the institutional (local) P53 IHC result.
6. Prior Therapy;

   * Naïve to first line systemic anti-cancer treatment. For patients with recurrent disease only, prior systemic anti-cancer treatment is allowed only if provided adjuvant chemotherapy was completed ≥ 12 months prior to randomization.

     a. Note : For Part A(Safety lead in phase), patient who used Paclitaxel, Carboplatin and Pembrolizumab for first line systemic therapy can participate if they meet all of the following conditions. Patient must have had 6 cycles of chemotherapy; patient must have physician assessed stable disease (SD), partial response (PR), or complete response (CR) after 6 cycles of therapy and patient must be enrolled within 9 weeks of their last dose of chemotherapy (last dose is the day of the last infusion)
   * Patients may have received prior radiation therapy for treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy. All radiation therapy must be completed at least 4 weeks prior to randomization.
   * Patients may have received prior hormonal therapy for treatment of endometrial cancer. All hormonal therapy must be discontinued at least three weeks prior to randomization.
7. Archival tumor tissue available or a fresh biopsy must be obtained prior to randomization.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
9. Have adequate organ function. Specimens must be collected within 7days prior to the start of study intervention.

   - Hematology Absolute neutrophil count (ANC) ≥1,500/μL without growth factor support within 2 weeks before screening test.

   Platelet ≥100,000/μL without transfusion within 2 weeks prior to screening test.

   Hemoglobin ≥10.0 g/dL without transfusion within 2 weeks prior to screening test.
   * Kidney function Creatinine or measured or calculated creatinine clearance (GFR may also be used in place of creatinine or CrCl a) ≤1.5 × ULN or ≥30 mL/min for subjects with creatinine levels >1.5 × institutional ULN.
   * liver function Total bilirubin ≤1.5×ULN or direct bilirubin ≤ULN for subjects whose total bilirubin exceeds 1.5 times the normal value.

   AST (SGOT) and ALT (SGPT) ≤3 × ULN (≤5 × ULN in subjects with liver metastases)
   * Coagulation International normalized ratio (INR) or prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5
   * Thyroid function Thyroid stimulating hormone (TSH) within normal limits (WNL); In euthyroid subjects receiving thyroid replacement therapy, TSH < ULN; If an abnormal TSH result is shown, free T4 is normal, and glandular function (euthyroid) is clinically normal, registration is possible.
10. Patient has voluntarily agreed to participate by giving written informed consent/assent for the trial.
11. Women of childbearing potential (WOCBP) must agree to use adequate contraception (hormonal method or abstinence, contraceptive procedure (IUD, Mirena, etc.)) from up to 14 days prior to randomization (for oral contraceptives), during treatment, and for 6 months after the last dose of Paclitaxel + Carboplatin, for 4 months after the last dose of Pembrolizumab, for 3 months after the last dose of Nesuparib, whichever occurs last.
12. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Patients will be considered of nonreproductive potential if they are either:

    * Postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women <45 years of age, a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient); OR
    * Have a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to randomization; OR Have a congenital or acquired condition that prevents childbearing.

Exclusion Criteria:

1. Patient has undergone prior treatment with a known PARP inhibitor.
2. Patient has a known hypersensitivity to nesuparib, pembrolizumab or combination cytotoxic chemotherapy components or excipients.
3. MMR deficiency confirmed by institutional MMR IHC testing.
4. Patients who are currently participating and receiving cancer-directed study therapy or have participated in a study of an investigational agent and received cancer-directed study therapy within 4 weeks prior to randomization.
5. Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with treated brain metastases may be eligible if follow-up brain imaging after CNS directed therapy shows no evidence of progression, and they have been off steroids for at least 4 weeks prior to randomization and remain clinically stable.
6. Patient has a known additional malignancy that progressed or required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
7. Patient has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
8. Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomization.

   * Patients who have received steroids as CT scan contrast premedication may be enrolled.
   * The use of inhaled or topical corticosteroids is allowed.
   * The use of mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
   * The use of physiologic doses of corticosteroids may be approved after consultation with the study chair.
9. Patients who have a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
10. Patient with uncontrolled intercurrent illness including, but not limited to: ongoing or active infection (except for uncomplicated urinary tract infection), interstitial lung disease or active, noninfectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
11. Patient has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
12. History of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as detectable HCV RNA [qualitative]) infection. Note: Testing for Hepatitis B or C is not required unless mandated by local health authority.
13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
14. Patient has known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
15. Patients with systemic autoimmune disease such as Systemic Lupus Erythematosus.
16. Has not adequately recovered from major surgery or has ongoing surgical complications.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding or expecting to be pregnant or conceive children within the projected duration of the study, starting with the screening visit through 6 months after the last dose of Paclitaxel + Carboplatin, 4 months after the last dose of Pembrolizumab, 3 months after the last dose of Nesuparib, whichever occurs last.
20. Has had an allogenic tissue/solid organ transplant.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | Assessed during 21days from day 1 of first combination maintenance treatment cycle (i.e., 21 days of Cycle 8 from day 1)
  In Part A, To evaluate dose-limiting toxicities(DLTs) of combination maintenance treatment with pembrolizumab and nesuparib during the 21 days from first nesuparib and pembrolizumab administration, and to establish a recommended Phase 2 dose(RP2D) and dosing schedule.
Overall distribution of progression-free survival | Approximately 11.01 months
  The time from randomization to the time when Progressive disease(PD) is first confirmed after administration of the first investigational drug (Pembrolizumab) or until death without disease progression.

SECONDARY OUTCOMES:
3, 6, 9 12-month Progression-free rate(PFS rate) | 3month, 6month, 9month, 12month after the study enrollment
  the proportion of patients who are alive and without disease progression after administering the investigational product
Median Progression-free time(Median PFS time) | All 36 subjects in each groups are enrolled and the 18-month follow-up period ends
  the proportion of patients who are alive and without disease progression after administering the investigational product
Overall response rate(ORR) | All 36 subjects in each groups are enrolled and the 18-month follow-up period ends
  the proportion of patients achieving complete remission(CR) or partial response(PR) as assessed by the Investigator per RECIST(v1.1) in patients who enter the study with measurable disease.
Duration control rate(DCR) | All 36 subjects in each groups are enrolled and the 18-month follow-up period ends
  the proportion of subjects who have achieved a best overall response of complete remission(CR), partial response(PR), or stable disesae(SD) per RECIST v.1.1 based on Investigator assessment.
Duration of response(DOR) | All 36 subjects in each groups are enrolled and the 18-month follow-up period ends
  DOR applies only to subjects whose BOR was CR or PR in patients who enter the study with measurable disease according to RECIST v.1.1 using the Investigator's tumor assessment. The start date is the date of first documented response (CR or PR), and the end date is the date defined as first documented PD or death due to any cause. If a subject had not had an event, duration will be censored at the date of last adequate tumor assessment.
Overall survival(OS) | All 36 subjects in each groups are enrolled and the 18-month follow-up period ends
  the time from the first date of investigational product administration to the date of death for any reason.
Progression free survival 2(PFS2) | All 36 subjects in each groups are enrolled and the 18-month follow-up period ends
  the time from the first date of administration of the investigational product to the earlier of disease progression or death in the subsequent anticancer therapy.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - National Cancer Center, Kyeonggi-do
  - Severance hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Kim SI, Cho HW, Choi CH, Park JY, Lee JB, Kim JW, Kim BG, Kim J, Lee JY. Phase II randomized study of first-line carboplatin and paclitaxel in combination with pembrolizumab, followed by maintenance pembrolizumab alone or with nesuparib, in mismatch-repair proficient, advanced or recurrent endometrial cancer (PENELOPE). J Gynecol Oncol. 2026 Jan;37(1):e50. doi: 10.3802/jgo.2026.37.e50. Epub 2025 Dec 22. PMID 41514313